CLINICAL TRIAL: NCT03104205
Title: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Home-Based Pilot
Brief Title: MOWI Home-Based Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John A. Batsis, MD, Associate Professor of Medicine and of The Dartmouth Institute Geisel School of Medicine at Dartmouth, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D16182_3; K23AG051681 (NIH)
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Results first posted 2021-12-20 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Obesity
Keywords: frail elderly; telemedicine; obesity; rural health; health promotion; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: A single arm pilot intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluate home-based MOWI (Experimental): Conduct and assess the feasibility, acceptability, and potential effectiveness of home-based MOWI in improving physical function.
  Interventions: Behavioral: Evaluate home-based MOWI

INTERVENTIONS:
Behavioral: Evaluate home-based MOWI — MOWI will be delivered via video-conferencing in the subject's home in a 3x per week, 26-week program from the coordinating center. It will include an individual dietician-led weekly nutrition session; 2x/week physical therapist-led group exercise session; and remote fitness device monitoring. We plan 5 cohorts of 8 subjects (n=40). In-person Research Assistant-led assessments will occur at 0, 8, 16 and 26 weeks. Recruitment, screening, selection criteria, and usability parallel Aim 2 (NCT03104192).

SUMMARY:
The goal of this study is to conduct a program of pilot research aimed at developing and evaluating a technology-assisted wellness intervention for older adults with obesity.

DETAILED DESCRIPTION:
The national epidemic of obesity is also affecting older adults, and is associated with an increased risk of disability, nursing home placement and early mortality. Conventional weight loss programs have the potential to reduce body fat, but are difficult to access for older obese adults due to transportation and mobility challenges. The overarching goal of this study is to conduct a program of pilot research aimed at developing and evaluating a technology assisted wellness intervention for older adults with obesity.

Study Timeline:

September 2018 to April 2021:

Goal: Conduct a study of improving weight and physical function in older adults with obesity at home using video-conferencing. An mHealth obesity wellness intervention (MOWI) will integrate a fitness device with a weekly individual dietician-led nutritional session, along with twice weekly physical therapist led group exercise session performed in a person's home.

Participation Duration: Three times weekly for 6 months. We shall also have participants return to the center once monthly

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Body Mass Index (BMI) ≥ 30kg/m^2 OR Waist circumference ≥88cm in females or ≥102cm in males
* Have Wi-Fi high speed internet
* Able to obtain medical clearance from doctor
* Have less than a 5% weight loss in past 6 months
* No advanced co-morbidity
* No exercise restrictions
* Not involved in other research studies that may interfere with participation

Exclusion Criteria:

* Severe mental or life-threatening illness
* Dementia
* Substance use
* History of bariatric surgery
* Suicidal ideation
* Unable to perform measures
* Reside in nursing home
* No advanced co-morbidity
* No exercise restrictions
* Not involved in other research studies that may interfere with participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Batsis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center / Dartmouth Medical School
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Batsis JA, Petersen CL, Clark MM, Cook SB, Kotz D, Gooding TL, Roderka MN, Al-Nimr RI, Pidgeon D, Haedrich A, Wright KC, Aquila C, Mackenzie TA. Feasibility and acceptability of a technology-based, rural weight management intervention in older adults with obesity. BMC Geriatr. 2021 Jan 12;21(1):44. doi: 10.1186/s12877-020-01978-x. PMID 33435877
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Amulet Technology Development & Validation — https://clinicaltrials.gov/show/NCT03085589
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Qualitative Assessment — https://clinicaltrials.gov/ct2/show/NCT03041831
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Research Pilot — https://clinicaltrials.gov/show/NCT03104192

RESULTS

PARTICIPANT FLOW:
Groups:
- MOWI Group: Single arm study that includes the cohort. There was one arm in this study of older adults with obesity that fulfilled criteria
Period: Overall Study
Arm/Group | MOWI Group
Started | 53
Completed | 44
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Evaluate Home-based MOWI
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in Grip Strength
Description: Assessed by a Jamar dynamometer. Sensor-based Thera-bands will measure data on strength change.
Time Frame: Change between baseline and follow-up at 26-weeks
Population: Evaluating those completing the intervention n=33. N=11 did not complete the follow-up evaluation as a result of COVID-19 restrictions.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MOWI Group
Number analyzed (Participants) | 33
kg | 1.2 (7.0)

2. Primary Outcome: Change in 30 Second Sit-to-Stand (STS)
Description: STS measures lower limb strength - change represented as repetitions.
Time Frame: Change between baseline and follow-up at 26-weeks
Population: Evaluating those completing the intervention n=44
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
repetitions | 3.1 (4.2)

3. Primary Outcome: Change in Six-Minute Walk Test (6MWT)
Description: A surrogate for cardiovascular fitness that measures distance (normal 400-700m) related to function. A clinically important difference is 50-55m
Time Frame: Change between baseline and follow-up at 26-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MOWI Group
Number analyzed (Participants) | 33
meters | 42.0 (77.3)

4. Primary Outcome: Change in Gait Speed (Meters Per Second)
Description: Gait speed is measured by the time it takes to walk 20 meters. Gait speed predicts disability and mortality (a significant change is considered 0.1 meters per second).
Time Frame: Change between baseline and follow-up at 26-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | MOWI Group
Number analyzed (Participants) | 33
meters per second | -0.34 (0.14)

5. Primary Outcome: Change in Late-Life Function and Disability Instrument (LLFDI)
Description: LLFDI consists of a 32-item function and 16-item disability (life-task) scales that correlate with gait speed and lower limb function. For this instrument we use only the 32-item function and scores are scaled. Minimum 0, Maximum 100. Higher scores indicate higher levels of function
Time Frame: Change between baseline and follow-up at 26-weeks
Population: Evaluating those completing the intervention n=44
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
units on a scale | 3.4 (4.7)

6. Secondary Outcome: Behavioral Activation (Patient Activation Measure)
Description: Patient Activation Measure (PAM) assesses knowledge, confidence and skill for managing health and grouped into 4 levels revealing insights into attitudes, motivators, behaviors & outcomes. Score ranges from 0 to 100, higher scores indicate higher activation.
Time Frame: baseline and follow-up at 26-weeks
Population: Subjective data is analyzed baseline and follow-up of participants n=53
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOWI Group
Number analyzed (Participants) | 53
score on a scale
  Baseline | 69.4 (12.1)
  26-weeks | 77.0 (14.6)

7. Secondary Outcome: Subjective Health Status (PROMIS)
Description: Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Short Form. PROMIS is a 10-item instrument capturing physical, mental and social aspects of quality of life having undergone quantitative appraisal and is non-proprietary. A score of 50 indicates the population mean with a standard deviation of 10. Higher scores indicate better health.
Time Frame: Change between baseline and follow-up at 26-weeks
Population: these are completers
Measure: Mean (Standard Deviation); unit: Change in the T score on a scale
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
Change in the T score on a scale
  Physical Function | 3.63 (4.89)
  Mental Function | 2.65 (5.70)

8. Secondary Outcome: Change in Weight in kg
Description: Change in weight in kg
Time Frame: Change between baseline and follow-up at 26-weeks
Population: Evaluating those completing the intervention n=44
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
kg | -4.6 (3.5)

9. Secondary Outcome: Change in Body Mass Index (BMI) in kg/m^2
Description: Change in body mass index (BMI) in kg/m^2
Time Frame: Change between baseline and follow-up at 26-weeks
Population: Evaluating those completing the intervention n=44
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
kg/m^2 | -1.8 (1.4)

10. Secondary Outcome: Change in Waist Circumference in cm
Description: Change in waist circumference in cm
Time Frame: Change between baseline and follow-up at 26-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | MOWI Group
Number analyzed (Participants) | 33
cm | -2.6 (5.4)

11. Secondary Outcome: Steps
Description: Fitibit will assess steps
Time Frame: Change between baseline and follow-up at 26-weeks
Population: Evaluating those completing the intervention n=44
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
steps | 4078 (3819)

12. Secondary Outcome: Community Healthy Activities Model Program for Seniors Physical Activity Questionnaire (CHAMPS) -
Description: CHAMPS is a self-reported tool in older adults that assesses activity levels and types. A change in score represents a change in the rates of participants in that specific category. A lower number (mean) represents a decrease in the proportion of individuals, while a positive change indicates an increase in the rate of persons. For caloric input, this continuous measure aligns with changes in calories based on activity type per week.
Time Frame: Change between baseline and follow-up at 26-weeks
Population: These are the completers of the intervention
Measure: Mean (Standard Deviation); unit: Kcal/week
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
Kcal/week
  low intensity caloric expenditure per week (ckal/week) | 312.69 (1323.67)
  moderate intensity caloric expenditure (Kcal/wk) | 5.05 (10.54)

13. Secondary Outcome: Community Healthy Activities Model Program for Seniors Physical Activity Questionnaire (CHAMPS) - Frequency Per Week
Description: as for outcome 12
Time Frame: Change between baseline and follow-up at 26-weeks
Population: These are the completers of the intervention
Measure: Mean (Standard Deviation); unit: exercise frequency per week
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
exercise frequency per week
  Not Exercising Frequency (frequency per week) | -2.93 (15.06)
  Low intensity frequency (frequency per week) | 2.36 (7.90)
  moderate intensity frequency (frequency per week) | 2.68 (5.30)

14. Secondary Outcome: Community Healthy Activities Model Program for Seniors Physical Activity Questionnaire (CHAMPS) - Hours Per Week
Description: as for outcome 12
Time Frame: Change between baseline and follow-up at 26-weeks
Population: These are the completers of the intervention
Measure: Mean (Standard Deviation); unit: exercise hours per week
Arm/Group | MOWI Group
Number analyzed (Participants) | 44
exercise hours per week
  Not exercise duration (hours per week) | -0.23 (11.16)
  low intensity duration (hours/week) | 1.64 (5.35)
  moderate intensity duration (hours per week) | 1.65 (4.45)

ADVERSE EVENTS:
Time Frame: 6 months - duration of the intervention
Arm/Group | MOWI Group
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 1/53
Other Adverse Events (participants affected / at risk) | 14/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOWI Group (N=53)
Atrial Fibrillation (Cardiac disorders) | 1 (1) — emergency room visit for atrial fibrillatino
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOWI Group (N=53)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 14 (14) — Shoulder, Knee, Kneck

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT03104205/Prot_SAP_ICF_000.pdf